CLINICAL TRIAL: NCT03781674
Title: Evaluation of the Role of 200 mg Versus 400mg Vaginal Progesterone in Prevention of Preterm Labor in Twin Gestation With Short Cervix: a Double-Blind Randomized Controlled Trial
Brief Title: Role of 200 mg Versus 400mg Vaginal Progesterone in Prevention of Preterm Labor in Twin Gestation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/194/18
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Twin; Pregnancy, Affecting Fetus or Newborn
Keywords: Preterm birth; Twin gestation; Vaginal progesterone
MeSH Terms: conditions — Premature Birth | interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: a double-blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: a double-blind randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- progesterone 400mg (Active Comparator): Women received vaginal progesterone suppositories in a dose of 400 mg(4 tablets) daily beginning at 18-22 weeks gestational age
  Interventions: Drug: progesterone 400mg
- progesterone 200mg plus placebo to progesterone 200 mg (Active Comparator): Women received vaginal progesterone suppositories in a dose of 200 mg(2 tablets) daily beginning at 18-22 weeks gestational age plus 2tablets placebo to vaginal progesterone
  Interventions: Drug: progesterone 200mg; Drug: placebo to progesterone 200mg
- placebo to progesterone 400 mg (Placebo Comparator): Women received 4 tablets placebo to vaginal progesterone suppositories
  Interventions: Drug: placebo to progesterone 200mg; Drug: placebo to progesterone 400mg

INTERVENTIONS:
Drug: progesterone 400mg — Women received vaginal progesterone suppositories in a dose of 400 mg daily beginning at 18-22 weeks gestational age
  Other Names: Active Comparator
  Arms: progesterone 400mg
Drug: progesterone 200mg — Women received vaginal progesterone suppositories in a dose of 200 mg daily beginning at 18-22 weeks gestational age
  Other Names: Active Comparator
  Arms: progesterone 200mg plus placebo to progesterone 200 mg
Drug: placebo to progesterone 200mg — Women received placebo to vaginal progesterone 200 mg suppositories in a dose of (2 tablets) daily beginning at 18-22 weeks gestational age
  Other Names: Placebo comparator
  Arms: placebo to progesterone 400 mg; progesterone 200mg plus placebo to progesterone 200 mg
Drug: placebo to progesterone 400mg — Women received placebo to vaginal progesterone 400 mg suppositories in a dose of (4 tablets) daily beginning at 18-22 weeks gestational age
  Other Names: placebo comparator
  Arms: placebo to progesterone 400 mg

SUMMARY:
The objective of the present study is to evaluate the effectiveness of two doses of vaginal progesterone(200mg versus400mg) and placebo in improving gestational age in twin pregnancy and its subsequent impact on perinatal outcome.

DETAILED DESCRIPTION:
The use of progesterone in the prevention of preterm birth(PTB) in both singleton and multiple pregnancies has been extensively investigated. Arguably, the use of progesterone is biologically plausible given that uterine quiescence is maintained throughout pregnancy by progesterone and progesterone receptor-mediated inhibition of inflammation, which causes suppression of the contractile genes. There is no benefit of universal vaginal progesterone to reduce PTB rates in multiple pregnancies. One meta-analysis showed a benefit in adverse perinatal outcome in a subgroup of women with a short cervix ≤25 mm, suggesting it may be useful in this group, but the numbers in the study were small and further research is needed. There appears to be no long-term harm caused to infants exposed to progesterone in utero. So the aim of the present study is to evaluate the effectiveness of two doses of vaginal progesterone(200mg versus400mg) and placebo in improving gestational age in twin pregnancy and its subsequent impact on perinatal outcome

ELIGIBILITY:
Inclusion Criteria:

* Women pregnant in dichorionic twins.
* Transvaginal sonographic cervical length is <25 mm at 18-22 weeks gestational age.
* No symptoms, signs or other risk factors for preterm labor.

Exclusion Criteria:

* Known allergy or contraindication (relative or absolute) to progesterone therapy.
* Monochorionic twins.
* Known major fetal structural or chromosomal abnormality.
* Intrauterine death of one fetus or death of both fetuses.
* Fetal reduction in the current pregnancy.
* Cervical cerclage in the current pregnancy.
* Medical conditions that may lead to preterm delivery.
* Rupture of membranes.
* Vaginal bleeding.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women pregnant in dichorionic twins.
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Preterm labor before 34 weeks gestations | Up to 34 weeks gestational age
  Number of patients delivered before 34 weeks gestations

SECONDARY OUTCOMES:
Neonatal respiratory distress syndrome | At birth
  Number of neonates develop respiratory distress syndrome

OTHER OUTCOMES:
Early neonatal death | One month after birth
  number of neonates died within one month from birth

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided